CLINICAL TRIAL: NCT01242540
Title: Brain Activation During Accommodation to Painful Stimulation With Functional Imaging of Pain
Brief Title: Brain Activation During Accommodation to Painful Stimulation With FMRI
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jim Ibinson, Clinical Instructor, University of Pittsburgh
Other Study IDs: PRO10020252
Record Dates: First submitted 2010-11-15; First posted 2010-11-17 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Pain
Keywords: Pain; Functional Magnetic Resonance Imaging
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Blood oxygen level dependant (BOLD) functional magnetic resonance imaging (FMRI) investigations of pain have provided substantial insight into the workings of the human brain. To date, however, the vast majority of studies have dealt with short painful stimulations. This work will expand the investigators knowledge of how longer stimulations are processed by comparing the activation pattern from a two minute painful stimulation with that of an 30-second painful stimulus. The investigators hypothesis that accommodation to the longer stimulation will be evident by either decreases in signal intensity in brain areas known to process pain, or by increasing activity in brain areas thought to be responsible for the modulation of painful perception.

DETAILED DESCRIPTION:
Background: Over the past 14 years, BOLD FMRI studies have non-invasively shown that pain activates a matrix of areas, but that this activation decays during stimulation, possibly reflecting the body's ability to "accommodate" to the stimulation. The majority of these use short applications of pain lasting 1 to 30 seconds. However, investigators are now using stimulations much longer than the periods that were typical a few years ago. The effect of signal decay on the activation maps generated by these longer tasks is not known. Because the signal change in many of the subcortical areas involved in pain processing is low, errors in analysis due to neglecting the signal decay may induce significant artifact.

Materials and Methods: Using transcutaneous electrical nerve stimulation, 20 healthy volunteers will experience two different painful stimulations: a repeating 30-second long stimulation and a constant 2 minute stimulation. The brain activity for each will be determined and compared. In addition, the signal decay during each painful stimulation will be quantified and compared.

Significance: Investigators are using longer stimulations periods in an attempt to understand how the brain processes "real- life" pain instead of the artificial on-off pattern of earlier studies. However, significant attention has not been paid to the possible effect of accommodation on the stimulus and how this may impact the activity pattern found. In addition, proof of activation of pain-control areas like the periaquaductal gray while inverse changes are occurring in pain-perceiving areas has not been sought. This study will address both of these issues with a single BOLD FMRI experiment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 50
* Right-handed
* Male or female
* Healthy individuals not taking any medication.

Exclusion Criteria:

* Pregnancy
* Diagnosed with any treated or untreated medical or neurological conditions
* Using any prescription drugs, including antidepressants, pain medications, sedative medications, blood pressure medications, seizure medications, or antipsychotics. Oral contraceptives are permitted
* Using any over-the-counter medications including aspirin, Tylenol, or herbal supplements
* Using any illicit substances
* Contraindications to magnetic resonance imaging.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects will come from the general surrounding community.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2010-11; Primary Completion 2011-06 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
To determine the areas of brain activity from a 2 minute long painful stimulation | After a 2 minute long painful stimulation

CONTACTS AND LOCATIONS:
Overall Officials: James W Ibinson, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Ibinson JW, Small RH, Algaze A, Roberts CJ, Clark DL, Schmalbrock P. Functional magnetic resonance imaging studies of pain: an investigation of signal decay during and across sessions. Anesthesiology. 2004 Oct;101(4):960-9. doi: 10.1097/00000542-200410000-00022. PMID 15448530
- [Background] Peyron R, Laurent B, Garcia-Larrea L. Functional imaging of brain responses to pain. A review and meta-analysis (2000). Neurophysiol Clin. 2000 Oct;30(5):263-88. doi: 10.1016/s0987-7053(00)00227-6. PMID 11126640
- [Background] Tracey I, Ploghaus A, Gati JS, Clare S, Smith S, Menon RS, Matthews PM. Imaging attentional modulation of pain in the periaqueductal gray in humans. J Neurosci. 2002 Apr 1;22(7):2748-52. doi: 10.1523/JNEUROSCI.22-07-02748.2002. PMID 11923440
- [Background] Seifert F, Bschorer K, De Col R, Filitz J, Peltz E, Koppert W, Maihofner C. Medial prefrontal cortex activity is predictive for hyperalgesia and pharmacological antihyperalgesia. J Neurosci. 2009 May 13;29(19):6167-75. doi: 10.1523/JNEUROSCI.4654-08.2009. PMID 19439594